CLINICAL TRIAL: NCT06850246
Title: Safety and Effectiveness of High Frequency Electrocautery for Abdominal Fat Reduction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Chengxin Li, Professor., Chinese PLA General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 03010240620
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-06

CONDITIONS: BMI

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- radiofrequency technology (Experimental): First, the frequency of 470 kHz was selected, and the CRT resistance probe was performed for deep fat management operation for 10 minutes, and then the CET capacitive mode 470 kHz was selected for superficial fat operation for 6 minutes. Then, select the 940 kHz frequency CET capacitance probe for epidermal tightening operation for 4 minutes. The temperature is set by the energy value. In CRT mode, the energy value is set to 70, and it can reach above 42 ℃ within one minute. In CET mode, the energy value setting is adjusted to 75. The operation mode is to gradually raise the temperature to the midline after partially increasing the temperature at the side of the waist. The technique is mainly to move in a circle and lift to the midline.
  Interventions: Device: treatment of radiofrequency technology
- Placebo (Placebo Comparator): Under the condition that the machine is not turned on, the treatment is performed in the same operation time, mode and treatment area of the treatment group.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: treatment of radiofrequency technology — When operating, first select 470 kHz frequency, CRT resistance probe for deep fat management operation for 10 minutes, and then select CET capacitance mode 470 kHz for superficial fat operation for 6 minutes. Then, select the 940 kHz frequency CET capacitance probe for epidermal tightening operation for 4 minutes. The temperature is set by the energy value. In CRT mode, the energy value is set to 70, and it can reach above 42 ℃ within one minute. In CET mode, the energy value setting is adjusted to 75. The operation mode is to gradually raise the temperature to the midline after partially increasing the temperature at the side of the waist. The technique is mainly to move in a circle and lift to the midline.
  Arms: radiofrequency technology
Device: Placebo — Under the condition that the machine is not turned on, the treatment is performed in the same operation time, mode, and treatment area of the treatment group.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the intervention of radiofrequency technology can help treat abdominal fat hypertrophy and skin laxity in adults. The main questions it aims to answer are

* Does radiofrequency technology lower the abdominal subcutaneous adipose tissue height by ultrasound measurement?
* Does radiofrequency technology improve abdominal circumference data and lower the number of times participants need to use a rescue inhaler.

Researchers will compare the treatment side to the non-treatment side to see if radiofrequency technology works to treat abdominal fat hypertrophy and skin laxity?

Participants will:

* Accept the treatment of radiofrequency technology every week for 10 weeks.
* Visit the clinic 1 month and 3 months after the treatment ends for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Age 18 to 65 years old (including 18 and 65 years old), male or female;
3. The body mass index (BMI) is in the range of 22 ~ 35 (kg/m2) (including the cut-off value);
4. Maintain a stable weight and lifestyle (including calorie intake and exercise) throughout the clinical study period and within 6 months after the end of the study;
5. Non-pregnant and breastfeeding women who have no pregnancy plan and voluntarily take effective contraceptive measures during the screening period and the whole trial period, and have no sperm or egg donation plan.

Exclusion Criteria:

1. Patients who gained or lost more than 2.5 kg of weight during the study;
2. Patients who have used weight loss drugs or participated in weight loss-related programs within 6 months of the start of the study;
3. Have received or are about to receive surgery or liposuction in the abdomen, or have received lipolytic drugs injected in the abdomen, or have received abdominoplasty or cryo lipolysis;
4. History of abdominal/waist-related trauma or scar;
5. Patients with excessive accumulation of abdominal skin affecting the operation;
6. Implantation of metal-related articles in the abdomen;
7. Patients suffering from severe systemic diseases that are life-threatening (such as cardiac insufficiency, renal insufficiency, etc.);
8. Those who are equipped with dentures, pacemakers, or other internal metal implants (such as metal IUD rings, etc.);
9. Local skin infection and open skin injury;
10. Have a history of eating disorder or eating disorder;
11. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Height of abdominal subcutaneous adipose tissue | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 (Week 1 after last treatment), Week 14 (Month 1 after last treatment), Week 22 (Month 3 after last treatment)
  Ultrasound (GE LogiQ P6 ultrasound system, 132 GE Healthcare, Wauwatosa, WI) was used to measure the height of abdominal subcutaneous adipose tissue at four positions below the left and right abdomen three times respectively. A mold plate was designed to fix the ultrasound probe, centered on the umbilicus, and symmetrically symmetrically. Areas A and B are horizontal measurement of ultrasonic probe, which are located above and below the left/right abdomen respectively, and areas C and D are vertical measurement of ultrasonic probe, which are located outside and inside respectively.Each measurement site was divided into three measurements and the average value was taken, and the overall average value of the three averages of each site was taken as the final value.

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No